CLINICAL TRIAL: NCT06494475
Title: A Randomised, Observer-Blind Trial to Evaluate the Immunogenicity, Safety, and Reactogenicity of a Group B Streptococcus Vaccine (GBS-NN/NN2) When 1 Dose is Administered Concomitantly With the Tdap Vaccine in Healthy-non Pregnant Women 18 to 49 Years of Age Compared to When Each Vaccine is Administered Alone
Brief Title: GBS-NN/NN2 (50 µg of Each Fusion Protein [GBS-NN and GBS-NN2] in Combination With 500 µg Aluminum as Alhydrogel®) Given With and Without the Tdap Vaccine in Healthy Non-pregnant Women 18 to 49 Years of Age
Status: Not yet recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Minervax ApS (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: MVX009; 2023-508563-73-00 (EU CTIS Number); U1111-1300-2150 (Other: Unique Trial Number)
Record Dates: First submitted 2024-07-02; First posted 2024-07-10 (Actual); Last update posted 2024-07-10 (Actual); Status verified 2024-07

CONDITIONS: Streptococcus Agalactiae Infection
Keywords: Immunology; Group B Streptococcus Vaccine; Streptococcus Agalactiae; Tdap
MeSH Terms: conditions — Streptococcal Infections | interventions — Boostrix

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Group 1 (coadministration [CA] Group/1 upper limb) (Experimental): Participants will receive a single placebo dose on Day 1. They will then receive two doses of the GBS-NN/NN2 vaccine on Days 29 and 57, respectively. The second dose on Day 57 will be administered in combination with the Tdap vaccine, with both injections given in the same upper limb.
  Interventions: Drug: GBS-NN/NN2 vaccine; Drug: Tdap vaccine; Drug: Placebo
- Group 2 (CA Group/2 upper limbs) (Experimental): Participants will receive a single placebo dose on Day 1 and two doses of the GBS NN/NN2 vaccine on Days 29 and 57, respectively. The second dose on Day 57 will be administered in combination with the Tdap vaccine, with the GBS-NN/NN2 injection in one upper limb and the Tdap injection in the other upper limb.
  Interventions: Drug: GBS-NN/NN2 vaccine; Drug: Tdap vaccine
- Group 3 (non-coadministration [NCA] Group/1 upper limb) (Experimental): Participants will receive two doses of the GBS NN/NN2 vaccine on Days 1 and 29, respectively. On Day 57, they will receive a single dose of the Tdap vaccine administered in combination with a placebo, with both injections (Tdap and placebo) given in the same upper limb.
  Interventions: Drug: GBS-NN/NN2 vaccine; Drug: Tdap vaccine; Drug: Placebo
- Group 4 (NCA Group/2 upper limbs) (Experimental): Participants will receive two doses of the GBS-NN/NN2 vaccine on Days 1 and 29, respectively. On Day 57, they will receive a single dose of the Tdap vaccine, administered in combination with a placebo. The Tdap vaccine will be injected in one upper limb and the placebo in the other upper limb.
  Interventions: Drug: GBS-NN/NN2 vaccine; Drug: Tdap vaccine; Drug: Placebo

INTERVENTIONS:
Drug: GBS-NN/NN2 vaccine — Intramuscular injection.
Drug: Tdap vaccine — Intramuscular injection.
  Other Names: Boostrix®
Drug: Placebo — Intramuscular injection.
  Arms: Group 1 (coadministration [CA] Group/1 upper limb); Group 3 (non-coadministration [NCA] Group/1 upper limb); Group 4 (NCA Group/2 upper limbs)

SUMMARY:
The main objectives of the study are to demonstrate the non-inferiority of the immune response induced by co administered GBS-NN/NN2 and tetanus, diphtheria, and acellular pertussis (Tdap) compared to the separate administration of GBS-NN/NN2 and Tdap, to evaluate the reactogenicity of GBS NN/NN2 when administered alone or in combination with Tdap, and to evaluate the safety of GBS-NN/NN2 when administered alone or in combination with Tdap in terms of serious adverse events (SAEs) and unsolicited adverse events (AEs).

ELIGIBILITY:
Inclusion Criteria:

* Women ≥18 to ≤49 years of age with a body mass index (BMI) of >17.5 to <40 kg/m2.
* Able to read, understand and capable of giving personal signed informed consent.
* Participants who are willing and able to comply with all trial procedures including completion of the electronic diary (eDiary) using their own personal mobile phone for 28 days after each dose.
* Healthy females at enrolment, as determined by medical history, physical examination, and clinical judgement of the investigator or participants with well controlled, well treated underlying conditions which will not impact the trial assessments.
* Women of childbearing potential must be:

  1. Documented to be surgically sterile or post-menopausal, or
  2. Willing to practice true abstinence throughout the trial and have a negative pregnancy test on Day 1, or
  3. Having same sex partners only, or
  4. Using at least one highly effective contraceptive measure, such as adequate hormonal method (eg, contraceptive implants, injectables, oral contraceptives) or non-hormonal methods (eg, intrauterine device, intrauterine hormone releasing system) throughout the trial and have a negative pregnancy test on Day 1.
* Expected to be available for the duration of the trial and who can be contacted by telephone during trial participation.

Exclusion Criteria:

* Pregnant women (positive urine pregnancy test on Day 1), women planning to become pregnant during the trial, and breastfeeding women.
* Women of childbearing potential not planning or willing to take adequate contraception (defined in inclusion criteria) from enrolment until 28 days after the last vaccination.
* Current or history of drug or alcohol abuse, as judged by the investigator.
* History of severe adverse reaction associated with a vaccine and/or severe allergic reaction (eg, anaphylaxis) to any component of GBS-NN/NN2 or any diphtheria toxoid-containing or CRM197-containing vaccine.
* History of microbiologically proven invasive disease caused by GBS, such as primary or secondary bacteriaemia, septic arthritis, endocarditis, prosthetic joint infection, necrotising myositis and fasciitis or pyelonephritis.
* Acute febrile illness, fever (temperature ≥38 degrees Celsius) before randomisation or an acute infection in the 7 days before screening and before the first dose.
* Bleeding diathesis or condition associated with prolonged bleeding that would, in the opinion of the investigator, contraindicate intramuscular injection.
* Any acute or chronic medical condition that, in the investigator's judgement, would make the participant unsuitable for participation in the trial.
* Any psychiatric condition, including recent (within the past year) active suicidal ideation/behaviour that may increase the risk of trial participation or, in the investigator's judgement, make the participant unsuitable for participation in the trial.
* Previous vaccination with any licensed or investigational GBS vaccine, or planned receipt during participation in the trial (from the first to the last visit).
* Vaccination within the previous 5 years with the Tdap vaccine or a vaccine containing any individual component thereof.
* Participants who have received any vaccine within 30 days of the first dose, or who are planning to receive any vaccine (eg, travel vaccines) up to 30 days after each dose and/or 7 days prior to the third dose.
* Participants who have received antipyretics/analgesics treatment within 72 hours prior to administration.
* Participants receiving immunosuppressive or immunomodulatory therapy, including steroids at immunosuppressive doses (10 mg or more prednisolone equivalent daily for 2 weeks or more during the past) or immunoglobulins in the 6 months prior to screening.
* Receipt or planned receipt of blood/plasma products, from 60 days before the first dose until the end of the trial.
* Participation in other trials involving investigational drug/vaccine(s) within 28 days prior to trial entry and/or planned during the trial.
* Participants with a deltoid muscle not being sufficiently large to permit the administration of 2 separate vaccinations at the same time visit, as determined by the investigator.
* Any personnel involved in the conduct of the trial (and their family members), including but not limited to, site staff members, MinervaX employees, and any vendor or contract research organisation (CRO) employees.

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 564 (Estimated)
Dates: Start 2024-12-17 (Estimated); Primary Completion 2025-06-21 (Estimated); Study Completion 2025-06-21 (Estimated)

PRIMARY OUTCOMES:
Number of Participants Expressing Anti-tetanus Toxoid Antibody Concentration ≥0.1 IU/mL | Day 85
Number of Participants Expressing Anti-diphtheria Toxoid Antibody Concentrations ≥0.1 IU/mL | Day 85
Number of Participants Expressing Anti-pertussis Toxin Antibodies | Day 85
Number of Participants Expressing Anti-filamentous Hemagglutinin (FHA) Antibodies | Day 85
Number of Participants Expressing Anti-pertactin (PRN) Antibodies | Day 85
Number of Participants Expressing RibN Antibody | Day 85
Number of Participants Expressing Alp1N Antibody | Day 85
Number of Participants Expressing Alp2N Antibody | Day 85
Number of Participants Expressing AlpCN Antibody | Day 85
Number of Participants Experiencing Solicited Local Adverse Events (AEs) | Day 63
Number of Participants Experiencing Solicited Systemic AEs | Day 63
Number of Participants Experiencing Unsolicited AEs | Day 85
Number of Participants Experiencing SAEs | Day 85
  An SAE is any occurrence that results in death, poses a life-threatening situation, necessitates inpatient hospitalization or the extension of an existing hospital stay, leads to persistent or significant disability or incapacity, involves a congenital anomaly or birth defect, or is considered an important medical event that, while not resulting in death, being life-threatening, or requiring hospitalization, still warrants serious concern.

SECONDARY OUTCOMES:
Number of Participants Experiencing Medically-attended Adverse Events (MAAEs) | Day 85
  A MAAE is defined as an AE that leads to an unscheduled visit to a health care professional.